CLINICAL TRIAL: NCT06693102
Title: Digital Intervention Targeting Cancer-related Cognitive Impairments
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 742333
Record Dates: First submitted 2024-11-13; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Cancer; Cognitive Impairment
Keywords: cancer survivors; cancer-related cognitive impairments; cognitive remediation; cognitive training; cognitive challenges
MeSH Terms: conditions — Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Masking Description: Participants are not randomized before all pre-assessment questionnaires and tests are completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital intervention targeting cancer related cognitive imapriments. (Experimental): Participants will undergo a digital intervention designed to address cognitive impairments. The program includes psychoeducation, cognitive training exercises, compensatory strategies, and cognitive restructuring. Weekly therapist support will be available via a chat function to provide guidance and feedback. Participants are encouraged to complete the intervention within a six-week timeframe.
  Interventions: Behavioral: Digital intervention targeting cancer-related cognitive impairments
- Crossword and sudoku tasks (Active Comparator): Participants will engage in crossword and Sudoku tasks, with a minimum recommended practice of 15 minutes per day over a six-week period.
  Interventions: Behavioral: Crossword and sudoku taks

INTERVENTIONS:
Behavioral: Digital intervention targeting cancer-related cognitive impairments — The intervention is developed using a person-centered approach and includes key components such as psychoeducation, cognitive training, compensatory strategy training, and cognitive restructuring exercises. Participants receive weekly remote support from a therapist and are encouraged to complete the program within a six-week period.
  Arms: Digital intervention targeting cancer related cognitive imapriments.
Behavioral: Crossword and sudoku taks — Participants receive crossword and sudoku tasks. They are encourraged to solve such tasks for a minimum of 15 minutes daily for six weeks.
  Arms: Crossword and sudoku tasks

SUMMARY:
Cognitive deficits are frequently reported following cancer treatment and can significantly impact daily functioning. These cognitive impairments often persist for years after cancer treatment. This study aimed to examine several aspects of a newly developed digital intervention designed to address cognitive impairments. Specifically, it focused on: (1) evaluating the preliminary effects of the intervention, (2) identifying predictors of treatment response, (3) assessing the feasibility of both the intervention and the study design, (4) gathering participant feedback on the intervention, and (5) testing the applicability of the Norwegian version of the Working Memory Questionnaire within this patient group.

DETAILED DESCRIPTION:
Many cancer survivors report cognitive challenges, including problems with concentration, attention, memory, processing speed, and executive functions. These cognitive impairments can persist for years after cancer treatment and are associated with reduced functioning at home and work.

Several approaches for managing cognitive difficulties are described in the literature. One approach is drill-and-practice interventions involving repetitive cognitive training, often employing computer-based tasks that increase in difficulty. Other interventions focus on strategy-based exercises, teaching patients to apply coping strategies in everyday situations. Additionally, psychoeducation is an important component in treating cognitive impairments.

Access to interventions for cognitive impairments remains limited. This limited may be a consequence of limited healthcare professionals resources. One potential solution is to offer digital interventions. The research literature shows that digital interventions are as effective as face-to-face treatment for mental health conditions such as anxiety and depression. In a previous study, we also found that digital interventions for cognitive impairments in depression, to be feasible. Offering digital interventions for cancer-related cognitive impairments might therefore be a promising approach for addressing one of the most common late effects following cancer treatment.

This study aims to assess the preliminary effects and the feasibility of a digital intervention for cancer-related cognitive impairments. Specifically, it aims to reduce self-reported cancer-related cognitive impairments. Additionally, we will examine whether the intervention increase performance on objectively measured cognitive tests. Other outcomes are rumination, life satisfaction, fatigue, depressive symptoms, and anxiety symptoms. Qualitative feedback from participants on their experience with the intervention will be used to refine the program. We will also assess the feasibility of a recently translated questionnaire for measuring working memory in this patient group. The study will include 60 cancer survivors. Thirty of these will receive the digital intervention and 30 will receive paper and pencil crossword and sudoku tasks.

The research questions are:

1. What preliminary changes in self-reported cognitive impairments and other clinical outcomes are observed among cancer survivors after receiving the digital intervention?
2. To what extent do clinical and demographic factors influence the usage and response to a digital intervention for cognitive impairments following cancer treatment?
3. How feasible is the newly developed digital intervention for cognitive impairments?
4. How do cancer survivors experience a newly developed digital intervention for cognitive impairments?
5. How effective is the translated version of the Working Memory Assessment Questionnaire in measuring cognitive impairments among Norwegian cancer survivors?

ELIGIBILITY:
The target group consists of individuals who have previously undergone cancer treatment (N=60).

Inclusion Criteria:

1. Age between 18 and 65 years,
2. Self-reported cognitive difficulties that are perceived to impact daily functioning (PCI <44 FACT-Cog),
3. Have received cancer treatment,
4. Completed curative treatment at least six months prior,
5. Proficient in speaking and writing Norwegian,
6. Access to a computer, tablet, or smartphone, and the internet.

Exclusion Criteria:

1. Neurological disorders (e.g., ADHD, MS, autism),
2. History of severe head injury,
3. Current moderate or severe depression (PHQ-9 score >14),
4. Previously diagnosed with serious mental disorders, such as substance abuse, bipolar disorder, or psychotic disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-02 (Estimated); Primary Completion 2028-01-02 (Estimated); Study Completion 2028-01-02 (Estimated)

PRIMARY OUTCOMES:
The Functional Assessment of Cancer Therapy- Cognitive Function | pre-assessment to two-year follow-up
  The Functional Assessment of Cancer Therapy- Cognitive Function (FACT-Cog) is a validated questionnaire consisting of 37 items designed to assess cognitive difficulties in cancer survivors. It includes four subscales: perceived cognitive impairment, cognitive abilities, feedback from others, and the impact of cognitive decline on quality of life. Total scores ranges from 0-148. Higher scores indicate better cognitive function.

SECONDARY OUTCOMES:
Digit Span Wechsler Adult Intelligence Scale-IV | Pre- to six-month follow-up assessments
  Digit Span Wechsler Adult Intelligence Scale-IV measures auditory attention span and working memory. Numbers are read aloud to participants, who repeat the sequence. The sequence length increases, and participants also repeat sequences backward. This test

OTHER OUTCOMES:
Rumination response scale | pre- to two year follow-up assessment
  Rumination response scale (RRS) consists of 22 items measuring aspects of rumination. Total scores ranges from 22-88. Higher scores indicate greater levels of rumination. The RRS can be divided into three subscales: depression-related thoughts, brooding, and reflection.
Patient Health Questionnaire-9 | Pre- to two-year follow-up assessment
  Patient Health Questionnaire-9 (PHQ-9) onsists of nine items that assess depressive symptoms. Scores ranges from 0-27. Higher scores indicate more symptoms. .
The Functional Assessment of Chronic Illness Therapy-Fatigue | Pre- to two years follow-up assessments
  The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT) is a 13-item questionnaire that assesses fatigue and its implications for daily functioning. Total scores ranges from 0 to 52. Higher scores represents less fatigue.
The Satisfaction with Life Scale | Pre-assessment to two-year follow-up
  The The Satisfaction with Life Scale (SWLS) measure life satisfaction. Total scores ranges from 5-35. Higher scores indicate greater level of life satisfaction. This questionnaire consists of five items.
Credibility and Expectancy Questionnaire | First week after receiving the intervention.
  The Credibility and Expectancy Questionnaire (CEQ) measure treatment credibility and expectancy. The rating scale ranges from 0-10 where higher scores indicate better credibility and expectancy.
California Verbal Learning Test II | Pre- to six-month follow-up assessments.
  The California Verbal Learning Test II (CVLT-II is a neuropsychological word list test measuring verbal short-term and long-term memory.
Color-Word Interference Test Delis-Kaplan Executive Function System | Pre- to six month follow-up assessments.
  The Color-Word Interference Test, from the Delis-Kaplan Executive Function System battery (D-KEFS), consists of four subtests. Two conditions measure processing speed and mental efficiency, where participants say the ink color of squares and read color names in black ink. The following conditions measure inhibition and focus-shifting, with one condition requiring participants to say the ink color of incongruent words, and the last requiring participants to switch between naming ink color and reading color words depending on whether a frame surrounds the word.
Word and Category Fluency Delis-Kaplan Executive Function System | Pre- six month follow-up assessments.
  The Word and Category Fluency, from the Delis-Kaplan Executive Function System (D-KEFS), is a neuropsychological test measuring verbal fluency. The test has three conditions: producing words that start with certain letters, naming items within categories, and alternating between categories.
The Generalized Anxiety Disorder-7 | Pre-assessment to two-year follow-up.
  The Generalized Anxiety Disorder-7 (GAD-7) consists of seven items that measure symptoms of anxiety. Total scores ranges from 0-21. Higher scores indicating more symptoms of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Anonymous data may be shared upon reasonable request, subject to restrictions imposed by data protection regulations.